CLINICAL TRIAL: NCT03761589
Title: Community-Academic Partnership to Promote Cardiovascular Health Among Underserved Children and Families
Brief Title: Efficacy of the Athletes for Life Program to Promote Cardiovascular Health
Acronym: AFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Noe Crespo, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14SDG20490382
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Fitness; Physical Activity
Keywords: Cardiovascular fitness; Physical Activity; Obesity; Children; Adults
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: Families (i.e., children and parents/primary caregivers dyads) were randomly assigned to participate in either the intervention group or a wait-list control group. The intervention (AFL) consisted of 24 structured, twice-weekly 90-min family-based, nutrition and sport/fitness-oriented sessions, and was delivered in a municipal recreation center. The wait-list control group received the intervention after all follow-up data had been collected. Data from all participants (both intervention group and wait-list group) were collected in four phases: before the intervention group started the program (week 0) and at 6, 12, and 24 weeks, thereafter.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AFL Intervention Group (Experimental): The AFL intervention consisted of twice a week physical activity and nutrition sessions for children and twice a week educational and physical activity sessions for parents. Each session lasted 90 minutes and all sessions were conducted in a municipal recreation center. The child program was delivered in English while the parent program was delivered in separate English-only or Spanish-only classes.
  Interventions: Behavioral: AFL Intervention
- Wait-List Control Group (Other): The wait-list control group received the 12-week AFL intervention after all follow-up data had been completed.
  Interventions: Behavioral: Wait-List Control

INTERVENTIONS:
Behavioral: AFL Intervention — The AFL intervention consisted of two 90-minute sessions per week for 12 months for both children and parents. The child physical activity sessions, held separately from the parent sessions, aimed to achieve 60 minutes of moderate-to-vigorous physical activity during each session through structured play activities, athletic drills, and sport exercises. Child dietary behaviors were taught through educational activities in small groups. For the parent program, behavior modification techniques were used to guide parents toward changing their own and their child's behavior. Take-home materials for self-monitoring of behaviors were used for both the child and the parent in order to reinforce concepts discussed in class.
  Arms: AFL Intervention Group
Behavioral: Wait-List Control — Families that were randomly assigned to the wait-list control group were asked not to change their normal physical activity or dietary behaviors for the duration of the 12-week waiting period. They were asked to participate in the baseline and 12-week evaluations and then they were enrolled to receive the 12-week intervention.
  Arms: Wait-List Control Group

SUMMARY:
The purpose of this study was to test the efficacy of a fitness- and behavioral-focused intervention, Athletes for Life (AFL), to improve cardiorespiratory fitness (CRF) among 160 underserved families.

DETAILED DESCRIPTION:
The Athletes for Life (AFL) study was a 12-week randomized controlled trial designed to promote cardiorespiratory fitness (CRF) and healthy lifestyle changes among parents and children. The original enrollment target was 160 families. A total of 149 parent-child dyads living in a Southwestern U.S. metropolitan area were enrolled in the study. AFL consisting of 24 structured, twice-weekly 90-min family-based, nutrition and sport/fitness-oriented sessions, and was delivered in a municipal recreation center. Behavior change, including increased physical activity, and adherence were motivated through positive reinforcement techniques. Families were randomized to either the AFL program or a wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Parent ages 18 years and over
* Child ages 6-11 years

Exclusion Criteria:

* Presence of a mental or physical condition that was contraindicated to participating in sports/exercise
* Having a chronic condition that limited mobility
* Taking medications that influenced body composition

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular fitness (total seconds) | 0, 12, and 24 weeks
  Child and adult cardiovascular fitness was assessed using a 1-mile run/walk test

SECONDARY OUTCOMES:
Change in insulin concentration (uIU/mL) | 0 and 12 weeks
  Child and adult insulin concentrations were measured via lipid panels and analyzed using Cobas automated analyzer.
Change in glucose concentration (mg/dL) | 0 and 12 weeks
  Child and adult glucose concentrations (plasma values) were measured via lipid panels and analyzed using Cobas automated analyzer.
Change in triglyceride concentrations (mg/dL) | 0 and 12 weeks
  Child and adult triglyceride concentrations were measured via lipid panels and analyzed using Cobas automated analyzer.
Change in total low-density lipoprotein (LDL) (mg/dL) | 0 and 12 weeks
  Child and adult LDL cholesterol values were measured via lipid panels and analyzed using Cobas automated analyzer.
Change in total high-density lipoprotein (HDL) (mg/dL) | 0 and 12 weeks
  Child and adult HDL cholesterol values were measured via lipid panels and analyzed using Cobas automated analyzer.
Change in average systolic blood pressure (mmHg) | 0, 12, and 24 weeks
  Child and adult systolic blood pressure was measured by an automated pressure cuff.
Change in average diastolic blood pressure (mmHg) | 0, 12, and 24 weeks
  Child and adult diastolic blood pressure was measured by an automated pressure cuff.
Change in total percent body fat (%) | 0, 12, and 24 weeks
  Child and adult percent body fat was measured via whole body Dual-energy X-ray absorptiometry (DXA) to assess body composition.
Change in total abdominal fat mass (g) | 0, 12, and 24 weeks
  Child and adult abdominal fat mass was measured via whole body Dual-energy X-ray absorptiometry (DXA) to assess body composition.
Change in total trunk percent fat (%) | 0, 12, and 24 weeks
  Child and adult trunk percent fat was measured via whole body Dual-energy X-ray absorptiometry (DXA) to assess body composition.
Change in waist circumference (inches) | 0, 12, and 24 weeks
  Child and adult waist circumference was measured via a tape measure.
Change in Body Mass Index (BMI) (kg/m^2) | 0, 12, and 24 weeks
  Child and adult BMI values were calculated using multiple measurements of height (cm) and weight (kg).
Frequency of fruit and vegetable consumption (times per month) | 0 and 12 weeks
  Child consumption of fruit and vegetables within the past month was measured via parental report using a Food Frequency Questionnaire (FFQ).
Frequency of dairy food consumption (times per month) | 0 and 12 weeks
  Child consumption of dairy foods (i.e., cheese, milk and yogurt) within the past month was measured via parental report using a Food Frequency Questionnaire (FFQ).
Frequency of protein consumption (times per month) | 0 and 12 weeks
  Child protein consumption (i.e., meat, fish, eggs and beans) within the past month was measured via parental report using a Food Frequency Questionnaire (FFQ).
Frequency of drink consumption (times per month) | 0 and 12 weeks
  Child consumption of drinks other than milk and 100% fruit juice (i.e., water, soda, and flavored drinks) within the past month was measured via parental report using a Food Frequency Questionnaire (FFQ).
Frequency of fat and sugar consumption (times per month) | 0 and 12 weeks
  Child consumption of fats and sugars (e.g., butter, potato chips, pastries) within the past month was measured via parental report using a Food Frequency Questionnaire (FFQ).
Frequency of grain consumption (times per month) | 0 and 12 weeks
  Child consumption of grains (e.g., cereals, brown rice, pasta) within the past month was measured via parental report using a Food Frequency Questionnaire (FFQ).
Change in physical activity (minutes per day of MVPA) | 12 weeks
  Child and adult 7-day physical activity (i.e., sedentary, moderate/vigorous activity) was measured using GENEActiv accelerometers.

CONTACTS AND LOCATIONS:
Overall Officials: Noe C Crespo, PhD, Principal Investigator — San Diego State University
Locations (1):
- Institute for Behavioral and Community Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szeszulski J, Vega-Lopez S, Todd M, Ray F, Behar A, Campbell M, Chavez A, Eckert R, Lorenzo-Quintero A, Hartmann Manrique L, Crespo NC. Athletes for life: Rationale and methodology of a community- and family-based randomized controlled trial to promote cardiovascular fitness among primarily Latino families. Contemp Clin Trials. 2020 Apr;91:105956. doi: 10.1016/j.cct.2020.105956. Epub 2020 Feb 13. PMID 32061969